CLINICAL TRIAL: NCT05089409
Title: A Phase 1, First in Human, Randomized, Double-Blind, Placebo-Controlled Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of ATB1651 in Adults With Mild to Moderate Onychomycosis
Brief Title: A Study of ATB1651 in Adults With Mild to Moderate Onychomycosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AmtixBio Co., Ltd. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ATB1651-101
Record Dates: First submitted 2021-10-12; First posted 2021-10-22 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A (ATB1651, 2 mg/mL) (Experimental): The planned ATB1651 dose level of 2 mg/mL.
  Six participants are expected to be enrolled in each arm.
  Interventions: Drug: ATB1651, 2 mg/mL
- B (ATB1651, 5 mg/mL) (Experimental): The planned ATB1651 dose level of 5 mg/mL.
  Six participants are expected to be enrolled in each arm.
  Interventions: Drug: ATB1651, 5 mg/mL
- C (ATB1651, 10 mg/mL) (Experimental): The planned ATB1651 dose level of 10 mg/mL.
  Six participants are expected to be enrolled in each arm.
  Interventions: Drug: ATB1651, 10 mg/mL
- D (ATB1651, 20 mg/mL) (Experimental): The planned ATB1651 dose level of 20 mg/mL.
  Six participants are expected to be enrolled in each arm.
  Interventions: Drug: ATB1651, 20 mg/mL
- E (ATB1651, 30 mg/mL) (Placebo Comparator): The planned ATB1651 dose level of 30 mg/mL.
  Six participants are expected to be enrolled in each arm.
  Interventions: Drug: ATB1651, 30 mg/mL
- F (placebo) (Placebo Comparator): The participants will apply placebo for 28 days.
  Six participants are expected to be enrolled in each arm.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ATB1651, 2 mg/mL — The participants will apply daily doses of ATB1651, 2 mg/mL to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: A (ATB1651, 2 mg/mL)
Drug: ATB1651, 5 mg/mL — The participants will apply daily doses of ATB1651, 5 mg/mL to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: B (ATB1651, 5 mg/mL)
Drug: ATB1651, 10 mg/mL — The participants will apply daily doses of ATB1651, 10 mg/mL to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: C (ATB1651, 10 mg/mL)
Drug: ATB1651, 20 mg/mL — The participants will apply daily doses of ATB1651, 20 mg/mL to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: D (ATB1651, 20 mg/mL)
Drug: ATB1651, 30 mg/mL — The participants will apply daily doses of ATB1651, 30 mg/mL to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: E (ATB1651, 30 mg/mL)
Other: Placebo — The participants will apply placebo to all 10 toenails including at least 1 affected great toenail for 28 days
  Arms: F (placebo)

SUMMARY:
The study is designed to evaluate the Safety, Tolerability and Pharmacokinetics of ATB1651 in participants with mild to moderate onychomycosis.

DETAILED DESCRIPTION:
Onychomycosis (also known as tinea unguium) is a contagious infection of toe nails by fungal organisms including dermatophytes, yeast, and molds.

This is phase 1, first in human, randomized, double-blind, placebo-controlled, MAD study designed to assess the safety, tolerability, and PK of ATB1651 when administered in participants with mild to moderate onychomycosis.

The study consists of 2 parts. In both parts, participants will receive multiple doses of ATB1651 applied to 1 affected great toenail and the remaining toenails (affected or not)

Part A: Participants will be enrolled into 1 of 3 cohorts and randomized to receive either ATB1651 or placebo at a ratio of 2:1.

Up to 2 additional cohorts may be added at the discretion of the Sponsor and Safety Monitoring Committee, if deemed necessary

Part B: Participants will be randomized within a single cohort to receive either ATB1651 or placebo at a ratio of 4:1

There will be 18 participants enrolled in part A, 30 participants in part B

ELIGIBILITY:
Inclusion Criteria:

1. Confirmation of onychomycosis by mycological staining and/or culture from affected great toenail(s).
2. Appearance of onychomycosis involving 20% to 70% of 1 (or both) affected great toenail(s) as determined by visual inspection after the nail has been trimmed. If the percentage of infection is outside this range but is still considered appropriate for this study, based on the overall impression of the Investigator, participation can be considered in consultation with the Medical Monitor.
3. The combined thickness of the distal nail plate at the associated hyperkeratotic nail bed is less than 3 mm.
4. Medically healthy with clinically insignificant Screening results (eg, laboratory profiles, medical history, ECGs, physical exam), as judged by the PI.
5. Negative urine drug screen and alcohol breath test at Screening and Day 1.
6. Body Mass Index (BMI) between 17.5 and 35.0, inclusive.
7. Agree to adhere to the current state and national advice regarding minimizing exposure to coronavirus disease of 2019 (COVID-19) from the Screening visit until the EOS visit.

Exclusion Criteria:

1. History of allergy to any of the excipients in ATB1651.
2. Positive COVID-19 test at Screening or any symptoms consistent with COVID-19 prior to initial dosing.
3. Positive test for hepatitis C antibody (HCV), hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody at Screening.
4. Have any underlying physical or psychological medical conditions that, in the opinion of the Investigator, would make it unlikely that the participant will comply with the study.
5. Pregnant or lactating at Screening or planning to become pregnant (self or partner) at any time during the study, including the follow-up period.
6. Unwilling to refrain from the use of nail cosmetics such as clear and/ or colored nail lacquers from the Screening visit until the end of the study.
7. Use of any IP or investigational medical device within 30 days prior to Screening, or 5 half-lives of the product (whichever is the longest) or participation in more than 4 investigational drug studies within 1 year prior to Screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple ascending doses (MAD) of ATB1651 in participants with mild to moderate onychomycosis through the percentage and severity of adverse events including pain, erythema and local irritation | From baseline to end of study treatment up to 56 days
  Adverse Events will be coded using the most current version of Medical Dictionary for Regulatory Activities (MedDRA®) Version 22.0 or higher

SECONDARY OUTCOMES:
To assess the efficacy of ATB1651 in improving signs and symptoms of onychomycosis in participants with mild to moderate onychomycosis | From baseline to end of study treatment up to 56 days
  Efficacy of ATB1651 assessed based on Mycological evaluation of the affected great toenail(s) where ATB1651 was applied
To assess the efficacy of ATB1651 in improving signs and symptoms of onychomycosis in participants with mild to moderate onychomycosis | From baseline to end of study treatment up to 56 days
  Difference in the appearance of the affected great toenail(s) as determined by photographs throughout treatment and follow-up periods
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Maximum plasma concentration and Time to maximum plasma concentration | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Apparent terminal elimination rate constant | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Area under the drug concentration-time curve, from time zero to 24 hours post dose | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Area under the drug concentration-time curve, from time zero to the last measurable concentration | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Area under the drug concentration-time curve, from time zero to infinity | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Apparent terminal half-life | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Apparent clearance | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Apparent terminal volume of distribution | From baseline to end of study treatment up to 56 days
To assess whether there is systemic exposure following multiple doses of ATB1651 through pharmacokinetic analysis Parameters: Plasma ATB1651 trough concentrations (Ctrough) during multiple dosing | From baseline to end of study treatment up to 56 days

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research Christchurch, Christchurch, New Zealand